CLINICAL TRIAL: NCT02630264
Title: A Randomized, Open-label, Multi-center Phase III Study Designed to Evaluate the Safety and Efficacy of E10A in Patients With Recurrent/Unresectable Squamous Cell Carcinoma of the Head and Neck Region
Brief Title: E10A for the Treatment of Squamous Cell Carcinoma of the Head and Neck
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Double Bioproducts Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E10AIII
Record Dates: First submitted 2013-12-26; First posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Head and Neck Neoplasms
Keywords: clinical trial; Recombinant Human Endostatin Adenovirus; randomized
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Endostatins; Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination therapy (Experimental): E10A+chemotherapy group (360 subjects):
  1. E10A (Endostatins) of 1.0×1012VP on day 1 and 6
  2. Paclitaxel Injection 160mg/m2 on day 3
  3. Cisplatin Injection 25mg/m2 on day 3, 4, and 5. Repeat every 21 days.
  Interventions: Drug: Endostatins; Drug: Paclitaxel injection; Drug: Cisplatin injection
- Chemotherapy (Experimental): Chemotherapy-alone group (180 subjects):
  1. Paclitaxel Injection 160mg/m2 on day 1
  2. Cisplatin Injection 25mg/m2 on day 1, 2, and 3. Repeat every 21 days
  Interventions: Drug: Paclitaxel injection; Drug: Cisplatin injection

INTERVENTIONS:
Drug: Endostatins — Specification: 1mL/division, 1×1012 VP/1.0mL
  E10A preparation:
  1. Thaw frozen E10A stored at -20°C vials at room temperature until E10A is liquid.
  2. Swirl gently. Do NOT shake.
  Method of administration
  1. E10A was diluted with 0.9% sodium chloride to appropriate dose according to the longest diameter of the target lesion.
  2. After local anesthesia, we penetrated the syringe under normal skin subcutaneously 5 mm into the tumor or vertically into the lymph node under direct visualization and withdrew it to confirm the absence of blood.
  3. Applied local compression for 10 minutes and pasted a sterile sticker on the injection site to avoid bleeding.
  Other Names: E10A
  Arms: Combination therapy
Drug: Paclitaxel injection — Specification:
  30mg/5mL,
  Usage:
  160mg/m2 on day 3, according to instruction.
Drug: Cisplatin injection — Specification:
  20mg
  Usage:
  Cisplatin 25mg/ m2 on day 3, 4, and 5,according to instruction.

SUMMARY:
Recombinant human endostatin adenovirus injection is a novel anti-tumor gene therapy drug. E10A contains a recombinant human endostatin gene with the second-generation recombinant adenovirus as its vector. After transfection tumor cells. E10A expresses human endostatin, which inhibits vascular endothelial cell proliferation and tumor angiogenesis, and blocks tumor blood supply, thereby specifically inhibiting tumor growth and inducing apoposis of tumor cells. Both pre-clinical and animal models have demonstrated the anti-tumor activities of E10A. The safety and efficacy of E10A in treating head and neck cancer has also been demonstrated in Phase I and Phase II studies.

DETAILED DESCRIPTION:
Phase II Clinical Study From March 2008 to December 2010 Safety and efficacy of intratumoral injections of E10A to cisplatin and paclitaxel was evaluated a multicenter, open-label, randomized clinical study in patients with advanced head and neck squamous cell carcinoma.

136 eligible patients were recruited and randomly assigned. Patients with locally advanced or metastatic head and neck squamous cell carcinoma or nasopharyngeal carcinoma not suitable for operation or radiotherapy were randomly assigned to receive E10A plus chemotherapy every 21 for a maximum of six cycles or to receive chemotherapy only.

The primary end point was the objective response rate (RR), defined as the proportion of patients who had a complete response (CR) or partial response (PR) at the target tumor lesion. The secondary end points were the objective disease control rate (DCR, or stable disease (SD) + PR + CR at the target tumor lesion), the overall RR, the overall DCR, OS, and progression-free survival (PFS).

The administration of E10A benefited some subgroups of patients. In the HNSCC patients, the objective RR was 36.5% (15/41) with E10A administration, exhibiting a trend of exceeding the rate of 20.0% (7/35) in the control group (P = 0.090; OR: 0.43), whereas the objective RR was 44.4% (12/27) versus 40.6% (13/32) in the NPC patients (P = 0.487; OR: 0.86). Patients who had previously received chemotherapy in the E10A group had a 44.8% (12/29) objective RR, whereas patients in the control group had only a 22.6% objective RR (7/31; P = 0.06, OR: 0.36). In contrast, patients without previous chemotherapy had a similar RR in both groups (34.3 versus 39.4%; P = 0.426, OR: 1.25).

The difference in the Kaplan-Meier estimates of PFS favored chemotherapy plus E10A, which resulted in a 3.43-month improvement. With a median follow-up of 10.47 months, the median PFS was 3.60 months (interquartile range: 2.60-7.63) in the control group and 7.03 months (interquartile range: 3.27-13.73) in the E10A group. As The median PFS was 3.60 months (interquartile range: 2.60-7.63) in the control group and 7.03months (interquartile range: 3.27-13.73) in the E10A group.

The OS of the E10A group was relatively prolonged in different subgroups compared with the controls (e.g., 13.37 months versus 9.67 months in the HNSCC patients, 13.03 months versus 10.50 months in those who had received prior treatment; Figure 1), but these results did not translate into significantly superior survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years with histologically or cytologically proven locoregionally advanced or metastatic HNSCC (excluding NPC) not suitable for operation or radiotherapy
2. A life expectancy≧12 weeks.
3. Patients were required to have at least one measurable (by imaging or photograph complied RECIST) lesion with the largest diameter ≧2 cm and suitable for the intratumoral injection of E10A,
4. Not received chemotherapy, radiotherapy, or biotherapy within 4 weeks.
5. Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0-2.
6. Adequate bone marrow,renal, and liver functions.

Exclusion Criteria:

1. Known allergies to the study drug.
2. The presence of important blood vessels/nerves or ulceration in the target lesion not suitable for injection.
3. Tumor relapses within 6 months after paclitaxel chemotherapy.
4. Severe coagulation disorders or bleeding tendency.
5. Severe uncontrolled medical conditions.
6. Recent history of myocardial infarction acute infection, pregnancy or lactation, or symptomatic brain metastases
7. A history of corticosteroids or immunosuppressives use within four weeks of study entry
8. Received any chemotherapy or radiotherapy within four weeks of study entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Time to progression | Up to 24 weeks
  Time to progression is defined as the time from randomization until objective tumor progression as verified for the first time

SECONDARY OUTCOMES:
Change in Overall response rate (CR+PR) | Up to 24 weeks, from date of randomization until the date of first documented progression
  the end of every 2 treatment cycles (each cycle is 21 days), and every 3 months during follow-up until disease progression. objective response rate (RR), defined as the proportion of patients who had a complete response (CR) or partial response (PR) at the target tumor lesion.
Chang in disease control rate (CR+PR+SD) | Up to 24 weeks, From date of randomization until the date of first documented progression
  the end of every 2 treatment cycles(each cycle is 21 days), and every 3 months during follow-up until disease progression.The CR or PR patients were reconfirmed
Incidence of Treatment-Emergent Adverse Events (Safety and tolerability) | Up to 32 weeks, from date of randomization until the date of first documented progression or date
  All adverse events were recorded regardless of their relevance to E10A
Overall survival | Up to 24 month, through study completion
  from cycle 2 to cycle 4 and calculated the survival during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Huiqiang Huang, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Guangzhou DB, Gaungzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ye W, Liu R, Pan C, Jiang W, Zhang L, Guan Z, Wu J, Ying X, Li L, Li S, Tan W, Zeng M, Kang T, Liu Q, Thomas GR, Huang M, Deng W, Huang W. Multicenter randomized phase 2 clinical trial of a recombinant human endostatin adenovirus in patients with advanced head and neck carcinoma. Mol Ther. 2014 Jun;22(6):1221-1229. doi: 10.1038/mt.2014.53. Epub 2014 Mar 25. PMID 24662947
- [Result] Lin X, Huang H, Li S, Li H, Li Y, Cao Y, Zhang D, Xia Y, Guo Y, Huang W, Jiang W. A phase I clinical trial of an adenovirus-mediated endostatin gene (E10A) in patients with solid tumors. Cancer Biol Ther. 2007 May;6(5):648-53. doi: 10.4161/cbt.6.5.4004. Epub 2007 Feb 13. PMID 17426445